CLINICAL TRIAL: NCT00268983
Title: A Multi-Center, Randomized, Phase 3 Study of Rituximab Versus Iodine I 131 Tositumomab Therapeutic Regimen For Patients With Relapsed Follicular Non-Hodgkins Lymphoma
Brief Title: Comparison Of Rituximab Versus Tositumomab and Iodine I 131 Tositumomab (BEXXAR® Therapeutic Regimen) For Patients With Relapsed Follicular Non-Hodgkins Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 393229/028
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Results first posted 2010-08-02 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: rituximab; tositumomab and iodine I 131 tositumomab; non-Hodgkins lymphoma; radioimmunotherapy; anti-B1 antibody; Bexxar; NHL; Tositumomab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tositumomab I-131; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tositumomab and Iodine I 131 Tositumomab (Experimental): Dosimetric dose: 450 mg Tositumomab infused over 1 hour followed by 5 mCi I 131 Tositumomab infused over 20 minutes
  Therapeutic dose: 450 mg Tositumomab infused over 1 hour followed by Individualized mCi activity of I 131 Tositumomab (35 mg) infused over 20 minutes.
  Interventions: Biological: Tositumomab and Iodine I 131 Tositumomab
- Rituximab (Active Comparator): Rituximab 375 mg/m2 given as an IV infusion once weekly for four weeks.
  Interventions: Biological: Rituximab

INTERVENTIONS:
Biological: Tositumomab and Iodine I 131 Tositumomab — Dosimetric dose: 450 mg Tositumomab infused over 1 hour followed by 5 mCi I 131 Tositumomab infused over 20 minutes
  Therapeutic dose: 450 mg Tositumomab infused over 1 hour followed by Individualized mCi activity of I 131 Tositumomab (35 mg) infused over 20 minutes.
  Other Names: Bexxar Therapeutic Regimen; anti-B1 Antibody; Iodine I 131 Tositumomab
  Arms: Tositumomab and Iodine I 131 Tositumomab
Biological: Rituximab — Rituximab 375 mg/m2 given as an IV infusion once weekly for four weeks.
  Arms: Rituximab

SUMMARY:
Comparison of rituximab versus Iodine I 131 Tositumomab Therapeutic Regimen (Tositumomab and Iodine I 131 Tositumomab or the Bexxar Therapeutic Regimen, formerly called Iodine-131 Anti-B1 Antibody) in subjects with follicular non Hodgkins B cell lymphoma. 506 subjects will be enrolled at 30 to 40 sites in the US, Canada, and Europe. Subjects will be randomly assigned to one of two treatment arms. In Arm A, subjects will receive 375 milligrams/meter2 (mg/m2 )of rituximab, given as an intravenous (IV) infusion once weekly for 4 weeks. In Arm B, subjects will undergo a two-phase treatment. In the first phase, termed the "dosimetric dose," subjects will receive an infusion of unlabeled Tositumomab (450 mg) immediately followed by an infusion of 5 millicuries (mCi) (0.18 gigabecquerel [GBq]) of Iodine 131 Tositumomab (35 mg). Whole body gamma camera scans will be obtained three times (Day 0; Day 2, 3, or 4; and Day 6 or 7) following the dosimetric dose. The information derived from the scans will enable a patient specific dose to be calculated to deliver the desired total body dose of radiation (65 or 75 centigray [cGy]). In the second phase, termed the "therapeutic dose," subjects in Arm B will receive an infusion of unlabeled Tositumomab (450 mg) immediately followed by an infusion of the subject specific activity of Iodine 131-conjugated Tositumomab (35 mg). Thyroid blockade will be implemented 24 hours prior to the dosimetric dose and continued for 14 days following the therapeutic dose. Subjects on study will be followed for response and safety at Week 7, Week 13, and every three months for the first and second year, every six months for the third year, and then annually for the forth and fifth years; and then for vital status, additional therapy, and long term safety events through year ten. Follow Up after subsequent NHL therapy will be carried out to assess tolerance of next anti-lymphoma therapy, development of myelodysplasia (MDS)/acute myelogenous leukemia (AML), HAMA or hypothyroidism, unexpected safety issues, and death.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed diagnosis of follicular lymphoma
* Recurrent lymphoma after one or two qualifying therapy regimen(s)
* Patients must not have progressed within 4 weeks of their last chemotherapy dose
* Rituximab may have been used once as a single agent, in one continuous course of 4-8 weekly infusions (10-week period), or in combination with chemotherapy in a single prior treatment
* Patients whose prior therapy includes rituximab must have had a 6 month or greater response duration following the rituximab-containing regimen.
* Performance status of at least 70% on the Karnofsky Scale and an anticipated survival of at least three months
* Adequate absolute neutrophil count and platelet count within 21 days of study entry without support of blood products/growth factors
* Adequate renal function and adequate hepatic within 21 days of study entry
* Measurable disease, with at least one lesion measuring >/=2.0 cm x 2.0 cm by CT scan
* Human Anti Mouse Antigen negative
* Written informed consent prior to study entry

Exclusion criteria:

* Histologic transformation to diffuse, large cell lymphoma.
* History of more than one course of Rituximab
* Disease limited to single lymph node or single group of nodes
* Involvement of 25% of the intratrabecular marrow by bone marrow biopsy specimen.
* Active infection requiring IV antibiotics at the time of study entry
* New York Heart Association Class III/IV heart disease
* Prior chemotherapy, biologic, radiation or steroid therapy for NHL within 8 weeks
* Any prior radioimmunotherapy
* Prior history of malignancy other than lymphoma (except for treated basal cell, squamous cell skin cancer, in situ cervical cancer, or other cancer that is disease-free for 5 years)
* Known HIV infection
* Hepatitis B positive
* Known central nervous system involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2004-10; Primary Completion 2009-09 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Walla Walla, Washington, United States
- GSK Investigational Site, Pierre-Bénite, France
- GSK Investigational Site, Manchester, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Quackenbush RC, Horner TJ, Williams VC, Giampietro P, Lin TS. Patients with relapsed follicular lymphoma treated with rituximab versus tositumomab and iodine I-131 tositumomab. Leuk Lymphoma. 2015 Mar;56(3):779-81. doi: 10.3109/10428194.2014.927461. Epub 2014 Jul 23. No abstract available. PMID 24898665
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 393229/028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 393229/028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 393229/028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 393229/028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 393229/028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 393229/028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 393229/028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study intended to recruit 506 participants to be randomized (1:1) to one of two treatment arms. However, due to feasibility issues, the study was stopped after only 15 participants were enrolled. Of these, 1 participant withdrew prior to receiving the first dose of study treatment; therefore, only 14 comprised the study population.
Groups:
- Rituximab 375 mg/m^2: Rituximab 375 milligrams per meters squared (mg/m^2) given as an intravenous infusion once weekly for four weeks (Day 0, Day 7, Day 14, and Day 21)
- TST/I-131 TST: Dosimetric dose, Given once on Day 1: Tositumomab (TST) infused over 1 hour, followed by 5 millicuries (mCi) I 131 Tositumomab (I-131 TST) infused over 20 minutes;
  Therapeutic dose, Given only once between Day 7 and Day 14:
  450 mg TST infused over 1 hour, followed by individualized mCi activity of I-131 TST (35 mg) infused over 20 minutes
Period: Overall Study
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Started | 6 | 8
Completed | 3 | 8
Not Completed | 3 | 0
Not completed — Death | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (14.4) | 53.1 (8.0) | 53.3 (11.0)
Gender [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 4 | 7
Race/Ethnicity, Customized [Number; unit: participants]
  White | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: Event-free survival is defined as the time from the date of randomization to the first occurrence of (whichever came first) progressive disease, death, or additional Non-Hodgkins Lymphoma (NHL) therapy due to disease-related symptoms, threatened end-organ function, cytopenias secondary to NHL, massive bulk disease, or steady progression over at least 6 months. Progressive disease is defined as at least a 50% increase in the sum of the perpendicular diameters of all measurable lesions and the appearance of new lesions at least 1.4 centimeters (cm) x 1.4 cm (i.e., 2.0 cm^2) by radiographic evaluation or greater than 1.0 cm by palpation upon physical examination.
Time Frame: From the date of randomization to the first occurrence of progressive disease, death, or additional Non-Hodgkins Lymphoma (median follow-up for the Rituximab and TST/I-131 TST groups was 62 and 91.5 months, respectively)
Population: Intent-to-Treat (ITT)-Exposed Population: all participants who received at least one dose of treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 6 | 8
Months | 9 [6.3 to 12.8] | NA [NA to NA] — Four of the 8 subjects in the TST/I-131 TST arm had not experienced an event by the time of their last follow-up, so there were insufficient events in the TST/I-131 TST arm to estimate the EFS, PFS or DOR

2. Primary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from the initial date of dosing to the first documented disease progression or death. Disease assessment was based on the International Workshop to Standardize Response Criteria (IWSRC) for Non-Hodgkin's Lymphoma (NHL). Progression is defined as at least a 50% increase in the sum of the perpendicular diameters of all measurable lesions and the appearance of new lesions at least 1.4 centimeters (cm) x 1.4 cm (i.e., 2.0 cm^2) by radiographic evaluation or greater than 1.0 cm by palpation upon physical examination.
Time Frame: From first dose of treatment until disease progression or death, whichever came first (median follow-up for the Rituximab and TST/I-131 TST groups was 62 and 91.5 months, respectively)
Population: ITT-Exposed Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 6 | 8
months | 9 [6.3 to 12.8] | NA [NA to NA] — Four of the 8 subjects in the TST/I-131 TST arm had not experienced an event by the time of their last follow-up, so there were insufficient events in the TST/I-131 TST arm to estimate the EFS, PFS or DOR

3. Secondary Outcome: Number of Participants Achieving Response
Description: Complete response (CR) is defined as the complete disappearance of all detectable clinical and radiographic evidence of disease and the disappearance of all disease-related symptoms (by the IWSRC) if present before therapy, and normalization of those biochemical abnormalities definitely assignable to NHL. Confirmation of response was carried out by an independent reviewer
Time Frame: Participants were followed for response at Week 7, Week 13, every 3 months for the first and second year, every 6 months for the third year, and then annually
Population: ITT-Exposed Population
Measure: Number; unit: Participants
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 6 | 8
Participants
  Complete response | 1 | 6
  Confirmed complete response | 1 | 6

4. Secondary Outcome: Duration of Response
Description: Response duration is defined as the time from the first documented response (complete response, complete response unconfirmed, or partial response) until disease progression. Partial response is defined as at least a 50% decrease in the product of two perpendicular diameters of all measurable lesions; no increase in the size of other nodes, liver, or spleen; and no new disease sites.
Time Frame: as for outcome 3
Population: ITT-Exposed Population. Only those participants with confirmed or unconfirmed complete response or partial response were analyzed for duration of response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 4 | 8
months | 7.3 [6.0 to NA] — The upper limit of the 95% confidence interval for the median was not estimable due to a small sample size and a small number of events. | NA [NA to NA] — Four of the 8 subjects in the TST/I-131 TST arm had not experienced an event by the time of their last follow-up, so there were insufficient events in the TST/I-131 TST arm to estimate the EFS, PFS or DOR

5. Secondary Outcome: Time to Death
Description: Time to death is defined as the time from treatment start to the date of death. As a median time to death is not presented for either group, see the outcome measure entitled "Number of Participants Who Had Died by the Month Indicated" for data regarding time to death.
Time Frame: as for outcome 2
Population: ITT-Exposed Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 6 | 8
months | NA [NA to NA] — Only 3 of the 6 subjects in the rituximab arm had died by the time of their last follow-up, so there were insufficient events to estimate median OS. | NA [NA to NA] — None of the 8 subjects in the TST/I-131 TST arm died by the time of their last follow-up, so there were insufficient events in the TST/I-131 TST arm to estimate median OS.

6. Secondary Outcome: Number of Participants Who Had Died by the Month Indicated
Description: The median time to death could not be calculated for participants in either treatment group; thus, data are shown as the number of participants who had died by the month indicated.
Time Frame: as for outcome 2
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 3 | 8
participants
  6.3 Months | 1 | 0
  33.1 Months | 1 | 0
  39.6 Months | 1 | 0

7. Secondary Outcome: Time to Next Treatment
Description: Time to next treatment is defined as time from the date of randomization until the new treatment is needed for NHL. Because too few evaluable participants were enrolled/treated, analysis of the time to next treatment was not conducted as planned.
Time Frame: Time from study randomization to 120 days after study drug administration
Population: ITT-Exposed Population
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Hematologic Nadir for Absolute Neutrophil Count
Description: Hematologic toxicity includes the analysis of hematologic nadir, which is defined as the lowest hematology value within 120 days of study drug administration.
Time Frame: Time from study randomization to 120 days after study drug administration
Population: ITT-Exposed Population excluding participants that did not have data within the 120 days of study drug administration.
Measure: Median (Full Range); unit: 10^3/cubic millimeter (mm^3)
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 0 | 3
10^3/cubic millimeter (mm^3) |  | 2.6 [1 to 4]

9. Secondary Outcome: Hematologic Nadir for Hemoglobin
Description: Hematologic nadir is defined as the lowest hematology value within 120 days of study drug administration.
Time Frame: Time from study randomization to 120 days after study drug administration
Population: ITT-Exposed Population
Measure: Median (Full Range); unit: Grams per deciliter (G/dL)
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 6 | 8
Grams per deciliter (G/dL) | 12.3 [10 to 15] | 11.6 [9 to 14]

10. Secondary Outcome: Hematologic Nadir for Platelet Count and White Blood Cell (WBC) Count
Description: Hematologic nadir is defined as the lowest hematology value within 120 days of study drug administration.
Time Frame: Time from study randomization to 120 days after study drug administration
Population: ITT-Exposed Population
Measure: Median (Full Range); unit: 10^3/microliter (µL)
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 6 | 8
10^3/microliter (µL)
  Platelets | 161.5 [138 to 324] | 57.0 [18 to 84]
  WBC Count | 4.8 [3 to 7] | 1.8 [1 to 4]

11. Secondary Outcome: Time to Nadir Values for the Indicated Hematological Parameters
Description: Hematologic nadir is defined as the lowest hematology value within 120 days of study drug administration. Time to nadir is defined as the number of days from the last administration of study drug to nadir.
Time Frame: Time from study randomization to 120 days after study drug administration
Population: ITT-Exposed Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 6 | 8
Days
  Absolute Neutrophil Count (n=0,3) | NA (NA) [NA to NA] — There was no participants available to determine absolute neutrophil count. | 17.0 (17.32)
  Hemoglobin (n=6,8) | 44.3 (25.57) | 38.5 (16.19)
  Platelet Count (n=6,8) | 33.3 (18.00) | 32.6 (4.21)
  WBC Count (n=6,8) | 45.8 (23.83) | 41.5 (4.93)

12. Secondary Outcome: Time to Recovery to Baseline Grade for the Indicated Hematological Parameters
Description: Hematologic nadir is defined as the lowest hematology value within 120 days of study drug administration. Time to recovery to Baseline grade is defined as the number of days from the last administration of study drug to a post-nadir hematology value of unmaintained Baseline grade or lower.
Time Frame: Time from study randomization to 120 days after study drug administration
Population: ITT-Exposed Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 6 | 8
Days
  Absolute Neutrophil Count (n=0,1) | NA [NA to NA] — There was no participants who had a drop in neutrophil count, therefore the Median and a 95% CI were unable to be calculated. | 7 [NA to NA] — There was only 1 participant with a baseline value ; therefore, time to recovery to baseline grade could only be evaluated for that one subject.
  Hemoglobin (n=6,8) | 46.5 [26.0 to 57.0] | 52.0 [29.0 to 77.0]
  Platelets Count (n=6,8) | 31.0 [22.0 to 57.0] | 49.5 [43.0 to 56.0]
  WBC Count (n=6,8) | 52.0 [28.0 to 64.0] | 73.0 [57.0 to 77.0]

13. Secondary Outcome: Duration of Grade 3/4 Toxicity for the Indicated Hematological Parameters
Description: Duration of Grade 3/4 toxicity is defined as the time between the date of the first Grade 3/4 lab result to the first lab date with a Grade of 0, 1, or 2 result. Laboratory abnormalities will be recorded as AEs using NCI CTCAE, Version 3, if they are associated with clinical squeal and/or require an intervention. Specific AEs not listed in the NCI criteria will be graded as follows: 1. Mild: An event that is easily tolerated by the subject, causing minimal discomfort and not interfering with everyday activities, 2. Moderate: An event that is sufficiently discomforting to interfere with normal everyday activities, 3. Severe: An event that prevents normal everyday activities, 4. Life-threatening or debilitating, and 5. Death
Time Frame: Time from study randomization to 120 days after study drug administration
Population: ITT-Exposed Population. Participants with a Grade 3/4 toxicity level for the indicated hematological parameters were analyzed (reflected by n=X, X). Different participants may have been analyzed for different parameters; thus, the overall number analyzed reflects everyone in the ITT-Exposed Population.
Measure: Median (Full Range); unit: Days
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 6 | 8
Days
  Absolute Neutrophil Count (n=0,1) | NA [NA to NA] — No participants reached Grade 3/4 toxicity so there was no duration to calculate. | 910 [910 to 910]
  Hemoglobin (n=0,0) | NA [NA to NA] — No participants reached Grade 3/4 toxicity so there was no duration to calculate. | NA [NA to NA] — No participants reached Grade 3/4 toxicity so there was no duration to calculate.
  Platelet Count (n=0,3) | NA [NA to NA] — No participants reached Grade 3/4 toxicity so there was no duration to calculate. | 22 [8 to 22]
  WBC Count (n=0,4) | NA [NA to NA] — No participants reached Grade 3/4 toxicity so there was no duration to calculate. | 22 [4 to 35]

14. Secondary Outcome: Number of Participants That Developed Hypothyroidism
Description: Hypothyroidism is defined as elevated Thyroid-Stimulating Hormone (TSH) or current history of using thyroid medication. The frequency of hypothyroidism at study enrollment will be determined, and participants with hypothyroidism at Baseline were excluded from analysis.
Time Frame: as for outcome 1
Population: ITT-Exposed Population
Measure: Number; unit: Participants
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 6 | 8
Participants | 0 | 2

15. Secondary Outcome: Number of Participants With an Infusion Reaction
Description: An infusion reaction is defined as any adverse event that occured within 24 hours of an infusion. An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Time Frame: First 24 hours of study drug administration.
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 6 | 8
participants | 0 | 1

16. Secondary Outcome: Number of Hospitalizations
Description: The frequency of hospitalizations within 90 days of treatment was summarized. Because too few evaluable participants were enrolled/treated, analysis of the number of hospitalizations was not conducted as planned.
Time Frame: Time of treatment until 90 days post-treatment
Population: ITT-Exposed Population
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Number of Participants With Myelodysplasia/Leukemia
Description: The cumulative incidence of myelodysplasia/leukemia was estimated.
Time Frame: as for outcome 1
Population: ITT-Exposed Population
Measure: Number; unit: Participants
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 6 | 8
Participants | 0 | 0

18. Secondary Outcome: Number of Participants With Any Serious Adverse Event (SAE) and Non-serious Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant temporally associated with the use of a medicinal product, whether or not it is considered related to the medicinal product. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is a Grade 4 (life threatening or disabling) non-hematologic laboratory abnormality assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: From randomization through Week 26
Population: ITT-Exposed Population
Measure: Number; unit: Participants
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Number analyzed (Participants) | 6 | 8
Participants
  Non Serious Adverse Evnts | 6 | 8
  Serious Adverse events | 4 | 4

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from randomization until Week 26 after participants' first dose. Beyond Week 26, events assessed as possibly related to study participation or drug administration were reported .
Arm/Group | Rituximab 375 mg/m^2 | TST/I-131 TST
Serious Adverse Events (participants affected / at risk) | 4/6 | 4/8
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 375 mg/m^2 (N=6) | TST/I-131 TST (N=8)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Peripheral T-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sebaceous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemorrhage (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 375 mg/m^2 (N=6) | TST/I-131 TST (N=8)
Headache (Nervous system disorders) | 2 | 5
Dizziness (Nervous system disorders) | 2 | 0
Dizziness postural (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1
Pyrexia (General disorders) | 3 | 1
Chills (General disorders) | 1 | 2
Fatigue (General disorders) | 1 | 2
Pain (General disorders) | 1 | 2
Application site rash (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Feeling cold (General disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Ligament disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 4
Lymphopenia (Blood and lymphatic system disorders) | 1 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 5
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 5
Vomiting (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Salivary duct obstruction (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 2 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 2
Breast mass (Reproductive system and breast disorders) | 1 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Euphoric mood (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Flushing: Vascular (Vascular disorders) | 2 | 0
Haemorrhage: Vascular (Vascular disorders) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 0 | 1
Venous pressure jugular increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Menopause (Social circumstances) | 0 | 1
White blood cells < 2000 cells/millimeters cubed (mm^3) (Investigations) | 0 | 4
Absolute neutrophill count < 1000 cells/mm^3 (Investigations) | 0 | 3
Platelets < 50000 cells/mm^3 (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.